CLINICAL TRIAL: NCT06621069
Title: The Effect of Long-term Use of Bisphosphonates on Femur Morphology
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0641
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Osteoporosis; Knee Osteoarthristis
Keywords: bisphosphonates; atypical femur fracture
MeSH Terms: conditions — Osteoporosis | interventions — Diphosphonates

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with over 5-year BP history: patients who took bisphosphonates over 5 years
  Interventions: Drug: Bisphosphonates
- control patients without BP usage: patients who do not receive bisphosphonates therapy
  Interventions: Other: Control

INTERVENTIONS:
Drug: Bisphosphonates — Alendronate Sodium or Zoledronic acid
  Groups: patients with over 5-year BP history
Other: Control — control without BP
  Groups: control patients without BP usage

SUMMARY:
Recent studies have shown that bone modeling can occur throughout life, suggesting bone has a persistent ability of adapting structure to loading. Some bone medications have a significant effect on the process of bone modeling based on histological studies. Bisphosphonates (BP), a classical anti-resorption drug which impacts the process of bone turnover, is related with atypical femur fractures while the mechanism is unclear. Several hypotheses are considered competitive. Among them, increased femur bowing is associated with atypical femoral fractures. However, it remains doubtful whether long-term BP use increases femur bowing. Thus, the investigators design this retrospective cohort study.

DETAILED DESCRIPTION:
If the participants meet the Inclusion Criteria, the investigators will collect the baseline characteristics of patients including age, gender, body mass index (BMI), as well as characteristics of BMD by dual-energy X-ray absorptiometry (DXA), BP treatment (type of drugs, duration before baseline). The primary outcome was femoral lateral bowing (FLB), femoral neck shaft angle (FNSA), and hip knee shaft angle (HKSA) from the frontal plane in standing radiographs of the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* standing radiographs of the lower limb

Exclusion Criteria:

* non-standard lower limbs X-ray , rheumatoid arthritis, tumor of the femur， congenital anomalies of the lower extremity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients are mostly from Zhejiang Province
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
femoral lateral bowing | through study completion, an average of 8 years
  Angle between axes of 20% proximal and distal sections of femur diaphysis

SECONDARY OUTCOMES:
femoral neck shaft angle (FNSA) | through study completion, an average of 8 year
  Angle between the femoral neck axis and mechanical axis of the femur
hip knee shaft angle | through study completion, an average of 8 years
  Angle between mechanical and anatomical femoral axes

CONTACTS AND LOCATIONS:
Locations (1):
- 1. Department of Orthopedics Surgery, The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China, Hangzhou, Zhejiang, China